CLINICAL TRIAL: NCT05883761
Title: Assessment of Birth Outcomes in Eswatini After Transition to Dolutegravir-based Treatment
Brief Title: Birth Outcomes In Eswatini After Transition To Dolutegravir-Based Treatment
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Ministry of Health Eswatini (Unknown); George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: EG0259
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-05

CONDITIONS: Neural Tube Defects; Congenital Abnormalities; Teratogens
MeSH Terms: conditions — Neural Tube Defects; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV-positive DTG preconception: HIV status defined as a documented positive result in the perinatal and/or maternity register or other clinical source record. Preconception drug exposure determined using date of DTG initiation and LMP date or gestational age at delivery (if LMP not available). ART at conception is defined as maternal ART that started up to 8 weeks after the calculated LMP date, which would be up to 6 weeks after the estimated date of conception. As this is the group of interest, sample size target was determined as 10,000.
- HIV-negative: Women with the last HIV test result recorded during pregnancy or labor and delivery as negative.
- HIV-positive on non-DTG ARV preconception: HIV status defined as a documented positive result in the perinatal and/or maternity register or other clinical source record. Preconception drug exposure determined using date of ARV initiation (e.g., efavirenz) and LMP date or gestational age at delivery (if LMP not available). ART at conception is defined as maternal ART that started up to 8 weeks after the calculated LMP date, which would be up to 6 weeks after the estimated date of conception. Other groups to be included as informed by the data (e.g., HIV+ not on ART a conception, unknown ART at conception, etc).

SUMMARY:
The goal of this observational study is to assess the birth outcomes of HIV-positive women delivering in hospitals in Eswatini who are receiving dolutegravir (DTG) or other anti-retroviral (ARV) drug regimens. The main question the study aims to answer is, what is the proportion of neural tube defects among live and stillborn infants delivered by:

* HIV-positive women on DTG at conception
* HIV-negative women
* HIV-positive women on non-DTG ARV at conception

Participants will be interviewed for information on HIV testing and antiretroviral therapy history, other medical history of selected conditions (e.g., diabetes, malaria, TB) and potential birth defect exposures. Photographs will be taken of the infants. Data on mothers' pregnancy history, birth outcomes, and HIV and ARV information (as applicable) will be collected from patient records.

DETAILED DESCRIPTION:
This is an observational study conducted at five high volume hospitals in Eswatini, in which birth defect and other data will be collected at the time of delivery (or hospital admission for miscarriages and medical abortions) for all women. The overall aim of this study is to evaluate the birth outcomes of HIV-positive women who are receiving DTG or other ARV drug regimens. The primary research objectives are to: 1) determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-positive women on DTG at conception; 2) determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-negative women; and 3) determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-positive women on non-DTG ART at conception. Secondary objectives are to determine overall general prevalence of major external birth defects and other pregnancy outcomes and any associations with other factors (e.g., maternal age, gravida). Data on mothers' pregnancy history, birth outcomes, and HIV and ARV information (as applicable) are collected from patient charts, registers, reporting forms and databases for all women. Women of live or stillborn infants with birth defects are consented for interviews capturing detailed history and exposure data and photographs of newborns' birth defects. Data collection will be for approximately 24 months. Blinded interview data and photographs are reviewed by a medical geneticist for confirmatory defect diagnosis. We will describe rates and 95% confidence intervals (CI) for birth defects among infants by maternal HIV and ART status.

ELIGIBILITY:
Surveillance component includes all deliveries/admissions as defined in study population description. For a subset of the population recruited for additional data collection:

Inclusion Criteria:

* women whose live or stillborn infant has birth defect as identified by a midwife or other clinician at the study hospital
* willing to provide informed consent

Exclusion Criteria:

* unable to provide informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women delivering infants at selected hospitals in Eswatini, including women delivering stillborn infants and those admitted for miscarriages or medical abortions due to identified congenital defects via diagnostic imaging
Sampling Method: Non-Probability Sample
Enrollment: 50075 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of neural tube defects (NTDs) among live and stillborn infants delivered by HIV-positive women on DTG at conception. | 24 months
  Number of live and stillborn infants with NTDs divided by the total number of live and stillborn infants of HIV-positive women on DTG at conception
Proportion of neural tube defects (NTDs) among live and stillborn infants delivered by HIV-negative women | 24 months
  Number of live and stillborn infants with NTDs divided by the total number of live and stillborn infants of HIV-negative women
Proportion of neural tube defects (NTDs) among live and stillborn infants delivered by HIV-positive women on non-DTG ARV at conception | 24 months
  Number of live and stillborn infants with NTDs divided by the total number of live and stillborn infants of HIV-positive women on non-DTG ARV at conception

SECONDARY OUTCOMES:
Prevalence of major external birth defects among all live and stillborn infants regardless of maternal HIV or ART status. | 24 months
  Number of live and stillborn infants with major external birth defects divided by the total number of live and stillborn infants among all women regardless of HIV or ART status
Proportion of other pregnancy outcomes | 24 months
  Number of live and stillborn infants with low birthweight and pre-term delivery divided by the total number of live infants among women (overall and by HIV/ART status); number of stillborn infants among all pregnancies, including miscarriages

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gill, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (5):
- Eswatini (5):
  - Good Shepherd Hospital, Lubombo, Lubombo Region
  - Hlathikhulu Hospital, Shiselweni, Shiselweni District
  - Mankayane Government Hospital, Manzini
  - Raleigh Fitkin Memorial Hospital, Manzini
  - Mbabane Government Hospital, Mbabane

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05883761/Prot_SAP_000.pdf